CLINICAL TRIAL: NCT04233840
Title: A Phase I/II Open Label Study to Evaluate Safety and the Prophylactic Effect on Recurrence of Anti-PD1 Monotherapy, P1101 Monotherapy, and Sequential Administration of P1101 and Anti-PD1 After Curative Surgery of HBV-related HCC
Brief Title: P1101 and Anti-PD1 for After Curative Surgery of Hepatitis B-related Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201710061MIPB
Record Dates: First submitted 2019-12-26; First posted 2020-01-18 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: P1101; Anti-PD1; HCC; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Phase I : Dose escalation study with Anti-PD1 dossages 4 cohorts Phase II : 3 parallel arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequential administration of P1101 and anti-PD1 (Experimental): Phase I of Study : To determine the safety, tolerability, DLT, and potential phase 2 dose of sequential administration of P1101 and anti-PD1
  :Sequential administration 6 doses (450mcg) of P1101 and 3 doses of anti-PD1 (Escalating from 0.3, 0.75, 1.5, 3 mg/kg) for Phase I Study
  Interventions: Drug: P1101 (Ropeginterferon alfa-2b); Drug: Nivolumab
- anti-PD1 (Active Comparator): Phase II Study Group I: anti-PD1 arm 3mg/kg 3 doses
  Interventions: Drug: Nivolumab
- P1101 monotherapy (Active Comparator): Phase II Study Group II: P1101 arm 450mcg 12 doses
  Interventions: Drug: P1101 (Ropeginterferon alfa-2b)
- sequential administration of P1101 and anti-PD1 (Experimental): Phase II Study GroupIII:Sequential administration of 6 doses of 450mcg P1101 and followed by 3 doses of anti-PD1 dosage (base on Phase I study result)
  Interventions: Drug: P1101 (Ropeginterferon alfa-2b); Drug: Nivolumab

INTERVENTIONS:
Drug: P1101 (Ropeginterferon alfa-2b) — solution for injection in prefilled syringe, 500 µg/ mL , 450μg /time, subcutaneous injection every 2 weeks
  Arms: P1101 monotherapy; Sequential administration of P1101 and anti-PD1; sequential administration of P1101 and anti-PD1
Drug: Nivolumab — Phase I study will use 0.3, 0.75, 1.5, 3mg/kg, Q2W for 3 doses after 6 doses of P1101.
  Phase II study : Group I will use 3mg/kg, Q2W for 3 doses; Group III will use the dosage that determine from Phase I study 3 doses after 6 doses of P1101
  Other Names: Opdivo
  Arms: Sequential administration of P1101 and anti-PD1; anti-PD1; sequential administration of P1101 and anti-PD1

SUMMARY:
The main purpose of this trial is to evaluate the safety of the new adjuvant treatment of curative HCC, or the treatment of long-acting interferon P1101 alone, or the use of long-acting interferon P1101 and subsequent treatment of anti-PD1, and any efficacy in reducing the recurrence rate of patients after surgery.

DETAILED DESCRIPTION:
secondary end-point: P1101 and anti-PD1 sequential therapy on hepatitis B (especially on HbsAg).

ELIGIBILITY:
Inclusion Criteria:

* Subject with HCC who meet the following criteria

  1. Subjects diagnosed as having typical HCC on dynamic CT, or dynamic MRI performed within 8 weeks before surgery, or subjects who diagnosed HCC by pathology after surgery resection;
  2. Subjects with the primary occurrence HCC ;
  3. Subjects with the HCC related to hepatitis B virus (HBV) ;
* Subject who have undergone surgical liver reaction within 8 weeks prior to study entry.
* Subjects showing a complete cure shows no findings suggestive of recurrence or remnant. ;
* Subject who are able to begin treatment with the study drug within 12 weeks after liver surgery resection. ;
* Subjects confirmed of satisfying the following conditions based on the screening performed at enrollment: Positive for HBsAg/ Undetectable HBV DNA, with or without current anti HBV treatment/ Grade A on Child-Pugh classification;
* Normal fundoscopic examination by ophthalmologist at screening;
* ECOG 0 to 1 ;

Exclusion Criteria:

* Subjects positive for anti-HCV ;
* Subjects showing vascular invasion of HCC on imaging diagnosis ;
* Subjects who have uncontrolled hypertension;
* Subjects with a history of pneumonitis or interstitial lung disease . cardiac arrest . an active infection requiring therapy .;
* Diabetes mellitus with HbA1c ≥ 7.4% with insulin treatment;

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Phase I portion - Dose-limiting Toxicity | 18 weeks
  To determine the potential phase 2 dose of sequestial administration of P1101 and anti-PD1. The MTD is determine by the prior dose level below the dose level at which ≥2/3 or ≥2/6 subjects suffer dose-limiting toxicity (DLT).
Phase II portion - Recurrence-free survival (defined as the time from randomization to HCC recurrence or death from any cause, whichever occured first) | 48 weeks
  To evaluate safety(assessment of AE, SAE and unanticipated problem) and the recurrence-free survival (defined as the time from randomization to HCC recurrence or death from any cause, whichever occured first) at 48 weeks after randomization of anti-PD 1 monotherapy, P1101 monotherapy, and sequential administration of P1101 and anti-PD 1 therapy arms

SECONDARY OUTCOMES:
Disease-free survival | 48 weeks
  To assess the effect of anti-PD1 monotherapy, P1101 monotherapy, and sequential administration of P1101 and anti-PD1 in inhibiting the recurrence, using disease-free survival (defined as the time from randomization to HCC recurrence, death from any cause, or onset of secondary tumor, whichever occurred first) at 48 weeks after randomization as the endpoint
Recurrence-free survival | 96 weeks
  To assess the treatment effect of anti-PD1 monotherapy, P1101 monotherapy, or sequential administration of P1101 and anti-PD1 in inhibiting the recurrence, using recurrence-free survival (defined as the time from randomization to HCC recurrence or death from any cause, whichever occurred first) at 96 weeks after randomization as the endpoint
HBsAg level | End of treatment of Anti-PD1 arm is up to 6 weeks; End of treatment of P1101 arm is up to 24 weeks; End of treatment of sequential administration of P1101 and anti-PD1 is up to 18 weeks, 24 weeks and 48 weeks
  To assess the change in mean HBsAg level from baseline at the end of treatment (EOT), 24 weeks and 48 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, Principal Investigator — NTUH
Locations (1):
- National Taiwan university Hospital, Taipei, Taiwan